CLINICAL TRIAL: NCT00934726
Title: Patient Satisfaction and Quality of Life Under Treatment With Seroquel XR
Brief Title: Non-interventional Open Label Study to Investigate the Effect of Quetiapine XR on Patient Satisfaction and Quality of Life in Patients With Schizophrenia
Acronym: PASQAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NAT-SER-2008/1
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Quality of Life in Schizophrenia
Keywords: Quality of Life; Patient satisfaction; Schizophrenia; Investigate quality of life in schizophrenia
MeSH Terms: conditions — Patient Satisfaction; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 group, schizophrenia patients: Patients with schizophrenia according to ICD-10(diagnostic and statistical manual of mental disorders)

SUMMARY:
Since subjective well-being and quality of life (QoL) are increasingly being recognized as important treatment outcomes in patients with schizophrenia (Hofer et al., 2004; Becker et al., 2005), the aim of this study is to investigate the effect of treatment with quetiapine XR on these parameters in the acute hospital and the subsequent ambulant care setting. The study is planned to be conducted in 15 centers all over Austria and, overall, about 150 inpatients with a ICD-10 diagnosis of acute schizophrenia are planning to be enrolled. The duration of the whole trial will be approximately 4 months, whereas 2 visits during hospitalization and two further visits after discharge will be scheduled. At each visit, adverse events and safety parameters, patient satisfaction and effectiveness of the current treatment, as well as concomitant medication and dosing schedules will be assessed and documented.In addition to that, the patients' overall satisfaction with antipsychotic therapy and their current quality of life will be determined using a QoL questionnaire, focussing on the subjective experience with quetiapine XR.

ELIGIBILITY:
Inclusion Criteria:

* Adult schizophrenia patients
* Inclusion according to Summary of product characteristics

Exclusion Criteria:

* Diagnosis other than schizophrenia
* Patients for which Seroquel XR is not registered (pregnant women, children and adolescents…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The psychiatrists according to inclusion criteria select patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Subject wellbeing under Neuroleptics scale (Quality of Life) | 4 months

SECONDARY OUTCOMES:
BPRS (Brief Psychiatric Rating Scale) | 4 months
CGI (Clinical Global Impression) | 4 months
All adverse events occurring during the study will be documented | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Siegfried Kasper, Prof., Principal Investigator — AKH Vienna